CLINICAL TRIAL: NCT02833701
Title: A Phase I Study of Bevacizumab and Intravenous Ascorbic Acid for Patients With Recurrent High Grade Glioma
Brief Title: Bevacizumab and Ascorbic Acid in Patients Treating With Recurrent High Grade Glioma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: University of Nebraska (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0769-15-FB; NCI-2016-00239 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P30CA036727 (NIH)
Record Dates: First submitted 2016-05-10; First posted 2016-07-14 (Estimated); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Glioblastoma; Glioma
MeSH Terms: conditions — Glioblastoma; Glioma | interventions — Ascorbic Acid; Bevacizumab; Immunoglobulin G; Disulfides

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (bevacizumab and ascorbic acid) (Experimental): Patients receive ascorbic acid IV over 90-120 minutes three times per week (at least 24 hours apart) and bevacizumab IV over 30-90 minutes on days 1 and 15. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Dietary Supplement: Ascorbic Acid; Biological: Bevacizumab; Other: Laboratory Biomarker Analysis; Other: Quality-of-Life Assessment

INTERVENTIONS:
Dietary Supplement: Ascorbic Acid — Given IV
  Other Names: 2-(1,2-dihydroxyethyl)-4,5-dihydroxy-furan-3-one; Asorbicap; C Vitamin; C-Long; Ce-Vi-Sol; Cecon; Cenolate; Cetane; Cevalin; L-Ascorbic Acid; VIT C; Vitamin C; Vitamin-C
Biological: Bevacizumab — Given intravenously (IV)
  Other Names: Anti-VEGF; Anti-VEGF Humanized Monoclonal Antibody; Anti-VEGF rhuMAb; Avastin; Bevacizumab Biosimilar BEVZ92; Bevacizumab Biosimilar BI 695502; Immunoglobulin G1 (Human-Mouse Monoclonal rhuMab-VEGF Gamma-Chain Anti-Human Vascular Endothelial Growth Factor), Disulfide With Human-Mouse Monoclonal rhuMab-VEGF Light Chain, Dimer; Recombinant Humanized Anti-VEGF Monoclonal Antibody; rhuMab-VEGF
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment

SUMMARY:
This phase I trial studies the side effects and best dose of ascorbic acid when given together with bevacizumab in treating patients with high grade glioma that has come back (recurrent). Monoclonal antibodies, such as bevacizumab may interfere with the ability of tumor cells to grow and spread. Ascorbic acid contains ingredients that may prevent or slow the growth of high grade glioma. Giving bevacizumab and ascorbic acid together may work better in treating patients with high grade glioma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the toxicities and determine the recommended dose of intravenous ascorbic acid given three times weekly in combination with intravenous bevacizumab every two weeks in patients with recurrent high grade glioma.

SECONDARY OBJECTIVES:

I. To evaluate changes in the levels of serum ascorbic acid (using high performance liquid chromatography [HPLC] with coulometric electrochemical detection) during therapy with ascorbic acid and bevacizumab.

II. Radiographic assessment of disease status after 2 cycles of therapy with ascorbic acid and bevacizumab.

III. To evaluate progression-free and overall survival of patients with recurrent high grade glioma treated with therapy with ascorbic acid and bevacizumab. Patients with stable or responsive disease after every 2 cycles will continue on therapy with ascorbic acid and bevacizumab until intolerance or progressive disease.

IV. To descriptively examine quality of life (QOL) using European Organization for Research and Treatment of Cancer (EORTC) Quality-of-Life Questionnaire QLQ-C30 during treatment.

OUTLINE: This is a dose-escalation study of ascorbic acid.

Patients receive ascorbic acid intravenously (IV) over 90-120 minutes three times per week (at least 24 hours apart) and bevacizumab IV over 30-90 minutes on days 1 and 15. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 2 months for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have pathologically proven diagnosis of high grade glioma
* Patients must have received prior radiation therapy and standard temozolomide; patients who have received additional therapies for previous progressions will be considered eligible
* Patients must be three or more months from the end of chemoradiotherapy or have biopsy or imaging consistent with disease progression
* Patients must have recovered from toxicity of prior therapy
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2 or better
* Absolute neutrophil count (ANC) >= 1,500/mm^3
* Hemoglobin >= 8 g/dL
* Platelet count >= 100,000/mm^3
* Serum creatinine that is at or below 2.0 mg/dL
* Serum aspartate transaminase (AST) and alanine transaminase (ALT) less than 1.5 times the upper limits of normal
* Serum alkaline phosphatase less than 2.5 times the upper limits of normal
* The patient must be aware of the neoplastic nature of his/her disease and willingly provide written, informed consent after being informed of the procedure to be followed, the experimental nature of the therapy, alternatives, potential benefits, side-effects, risks, and discomforts
* Women of reproductive potential must be non-pregnant and non-nursing and must agree to employ an effective barrier method of birth control throughout the study and for up to 6 months following treatment
* Women of child-bearing potential must have a negative pregnancy test within 7 days of initiating study; (no childbearing potential is defined as age 55 years or older and no menses for two years or any age with surgical removal of the uterus and/or both ovaries)

Exclusion Criteria:

* History of uncontrollable allergic reactions to bevacizumab or ascorbic acid
* Known human immunodeficiency virus (HIV)-positivity AND actively being treated with highly active antiretroviral therapy (HAART)
* History of glucose-6-phosphate dehydrogenase deficiency
* History of oxalate nephrolithiasis or urine oxalate >60 mg/dL
* Anuria, dehydration, severe pulmonary congestion or pulmonary edema or fixed low cardiac input
* Prior hypersensitivity to bevacizumab or toxicity requiring discontinuation of bevacizumab
* Clinically significant cardiovascular disease defined as follows:

  * Inadequately controlled hypertension (i.e., systolic blood pressure [SBP] > 160 mm Hg and/or diastolic pressure [DBP] > 90 mm Hg despite antihypertensive therapy)
  * History of cerebrovascular accident (CVA) within 6 months
  * Myocardial infarction or unstable angina within 6 months
* Evidence or history of bleeding diathesis (greater than normal risk of bleeding, i.e., Hereditary Hemorrhagic Telangiectasia type I or HHT-1) or coagulopathy in the absence of therapeutic anti-coagulation or any hemorrhage/bleeding event > grade 3 within 4 weeks prior to registration; note: patients with full-dose anticoagulants are eligible provided the patient has been on a stable dose for at least 2 weeks of low molecular weight heparin; therapeutic Coumadin and aspirin doses > 325 mg daily are not allowed
* Active wound, a serious or non-healing wound, an active ulcer or untreated bone fracture
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess =< 6 months prior to registration
* Major surgical procedure, open biopsy or significant traumatic injury =< 28 days prior to registration
* Any other clinically significant medical disease or condition laboratory abnormality or psychiatric illness that, in the Investigator's opinion, may interfere with protocol adherence or a subject's ability to give informed consent
* Patients who are on the following drugs and cannot have a drug substitution: flecainide, methadone, amphetamines, quinidine, and chlorpropamide; Note: high dose ascorbic acid may affect urine acidification and, as a result, may affect clearance rates of these drugs
* Simultaneous participation in other therapeutic clinical trials will not be allowed
* Inability to co-operate with the requirements of the protocol
* Pregnant and nursing women are excluded from this study

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2016-03; Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Frequency of occurrence of overall toxicity | Up to 52 weeks
  Categorized by toxicity grades
Incidence of dose limiting toxicities (DLT) | Up to 56 days
  Described by dose level
Incidence rates of adverse events | Up to 52 weeks
  Described by dose level
Maximum tolerated dose of ascorbic acid combined with bevacizumab | Up to 56 days
  Maximum tolerated dose of ascorbic acid in combination with bevacizumab defined as the highest dose tested which results in DLT in no more than 1 of 6 evaluable patients

SECONDARY OUTCOMES:
Changes in serum levels of ascorbic acid using HPLC with coulometric electrochemical detection | Week 1 to up to Week 52
  Correlation of intracellular glutathione with ascorbic acid levels during therapy with ascorbic acid and temozolomide will be summarized using descriptive statistics to summarize changes over time.
Disease status by radiologic assessment | Up to 56 days
  Disease status measured by radiologic assessment
Progression free survival | First date of therapy until the first notation of clinical progression, relapse or death from any cause, assessed up to 1 year
  Will be plotted following the method of Kaplan and Meier
QOL using EORTC QLQ-C30 | Up to 52 weeks
  Will be descriptively summarized using means and standard deviations.
Survival | First date of therapy until the date of death from any cause, assessed up to 1 year
  Will be plotted following the method of Kaplan and Meier.

CONTACTS AND LOCATIONS:
Overall Officials: Nicole A Shonka, MD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States